CLINICAL TRIAL: NCT03177551
Title: Development and Validation of Predictive Nomogram for Castration Resistant to Androgen Deprivation Therapy in Patients With Advanced Prostate Cancer
Brief Title: Predictive Nomogram of CRPC
Acronym: CRPC-PN
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tianjin Medical University Second Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CRPC-PN
Record Dates: First submitted 2017-05-31; First posted 2017-06-06 (Actual); Last update posted 2018-10-01 (Actual); Status verified 2018-09

CONDITIONS: Castration-resistant Prostate Cancer; Metastatic Cancer
Keywords: Prostatic Neoplasms; Nomograms; Drug Resistance, Neoplasm
MeSH Terms: conditions — Neoplasm Metastasis; Prostatic Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Developement Cohort: Development the Predictive Nomogram for mCRPC in Patients with Prostate Cancer
- Validation Cohort: Validation the Predictive Nomogram for mCRPC in Patients with Prostate Cancer

SUMMARY:
This is an observational, prospective (study following participants forward in time), multi-center (study conducted in more than 1 center) study to identify the risk factors, then develop and validate the predictive Nomogram of metastatic castration-resistant prostate cancer (mCRPC) that will effectively predict the early onset mCRPC in patients receiving androgen-deprivation therapy (ADT). The entire duration of study will be approximately 3 year. Participants will primarily be evaluated for achieving biochemical or radiological progression after receiving ADT based on EAU 2017 practice guideline criteria. Serum testosterone, prostate specific antigen (PSA), alkaline phosphatase (ALP) and blood routine will be monitored throughout the study.

DETAILED DESCRIPTION:
This is an observational, prospective (study following participants forward in time), multi-center (study conducted in more than 1 center) study to identify the risk factors, then develop and validate the predictive Nomogram of metastatic castration-resistant prostate cancer (mCRPC) that will effectively predict the early onset mCRPC in patients receiving androgen-deprivation therapy (ADT). The entire duration of study will be approximately 3 year. Participants will primarily be evaluated for achieving biochemical or radiological progression after receiving ADT based on EAU 2017 practice guideline criteria. Serum testosterone, prostate specific antigen (PSA), alkaline phosphatase (ALP) and blood routine will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants who have given consent form;
* Participants with pathologically defined prostate cancer;
* Participants with life expectancy of at least 6 months based on the Investigator's clinical judgment;
* Participants having indication and planning to receiving ADT.

Exclusion Criteria:

* Participants with previous history of ADT;
* Participants who are allergic to contrast medium;
* Participants who failed to regulate endocrine therapy with the orders requirements;

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male only
Study Population: Participants having indication and planning to receiving ADT.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2017-05-04 (Actual); Primary Completion 2019-09 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
Time to castration resistant | 3 YEARS
  The definition mCRPC is that the castrated androgen < 50 ng/dL or 1.7 nmol/L plus either;
  1. Biochemical progression: Three consecutive rises in PSA one week apart resulting in two 50% increases over the nadir, and a PSA > 2 ng/mL or,
  2. Radiological progression: The appearance of new lesions: either two or more new bone lesions on bone scan or a soft tissue lesion using RECIST (Response Evaluation Criteria in Solid Tumours) [736].
  Symptomatic progression alone must be questioned and subject to further investigation.

CONTACTS AND LOCATIONS:
Overall Officials: Yuanjie Niu, MD,PhD, Principal Investigator — Tianjin Medical University Second Hospital
Locations (1):
- Tianjin Medical Unversity Second Hospital, Tianjin, China

IPD SHARING:
Plan to Share IPD: Yes
IPD could be got by contacting researchers.